CLINICAL TRIAL: NCT03955133
Title: Polypharmacy and Adverse Drug Reactions: Nurse-led Intervention to Minimise Adverse Drug Reactions for Older Adults in Care Homes: a Quality Improvement Process Intervention
Brief Title: The Adverse Drug Reaction (ADRe) Profile for Polypharmacy
Acronym: ADRe-p
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Aneurin Bevan University Health Board (Other); Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SwanseaNursing
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2020-02

CONDITIONS: Polypharmacy
Keywords: medicines management; adverse drug reaction; care homes; nurses
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Polypharmacy

STUDY DESIGN:
Intervention Model Description: All participating care homes will receive the intervention at the same time. Residents' records and medicines charts will be reviewed sequentially.
Masking Description: Use of the intervention could not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): This is a single arm before and after study with data collection at 4 time points.
  Interventions: Other: Adverse Drug Reaction ADRe Profile for Polypharmacy

INTERVENTIONS:
Other: Adverse Drug Reaction ADRe Profile for Polypharmacy — PADRe asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the British National Formulary (BNF) and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts. A full description is published (references below).

SUMMARY:
Polypharmacy, the use of multiple or inappropriate medications, has the potential to harm older adults by causing cognitive impairment, falls, and hospitalisations. The nurse-led intervention (The ADRe Profile) to review mental health medicines has demonstrated improved care quality by: identifying serious adverse drug reactions (ADRs); reducing prescription of mental health medicines; reducing the prevalence of pain and nausea; and, increasing non-urgent national health service (NHS) contacts. The investigators will develop ADRe to encompass medicines commonly prescribed in primary care and evaluate intervention implementation in care homes in Aneurin Bevan University Health Board.

DETAILED DESCRIPTION:
The investigators will introduce medicines' monitoring using the PADRe Profile into up to 7 care homes, each with up to 26 residents prescribed >4 medicines (estimated ~90% residents).

Each home will identify a nurse lead and a deputy. Nurses will be asked to administer the PADRe Profile with all patients prescribed >4 medicines.

Barriers, facilitators, and feasibility of the Profile will be explored. This will identify how, in which contexts medicines' monitoring can be integrated into routine care, relate the Profile to improved processes and outcomes of care, and inform implementation strategies (see logic model in cited papers).

Data collection:

* Record review before and after each of 3 administrations of the intervention to identify clinical and prescription changes. Narrative accounts of problems causing moderate or severe harm will be prepared.
* Serial interviews and debriefs with nurses: three per nurse.
* Stakeholder interviews with patients, participating pharmacists and prescribers for an overview of implementation.

ELIGIBILITY:
Inclusion Criteria:

* • Resident at the care home and expected to continue to live there for 1 year

  * Currently taking >3 prescribed medicines daily
  * Willing and able to give informed, signed consent themselves, or where capacity is lacking, a consultee is willing to give advice and assent to the resident participating.

Exclusion Criteria:

* age <18

  * Prescribed <4 medicines daily;
  * Receiving active palliative care
  * Not well enough to participate, as screened by their nurses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sue jordan, PhD, Study Chair — Swansea University
Locations (1):
- Swansea University, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The terms of our ethical approval would not allow this.

REFERENCES:
- [Background] Jordan S, Logan PA, Panes G, Vaismoradi M, Hughes D. Adverse Drug Reactions, Power, Harm Reduction, Regulation and the ADRe Profiles. Pharmacy (Basel). 2018 Sep 18;6(3):102. doi: 10.3390/pharmacy6030102. PMID 30231573
- [Background] Jordan S, Banner T, Gabe-Walters M, Mikhail JM, Round J, Snelgrove S, Storey M, Wilson D, Hughes D; Medicines Management Group. Nurse-led medicines' monitoring in care homes study protocol: a process evaluation of the impact and sustainability of the adverse drug reaction (ADRe) profile for mental health medicines. BMJ Open. 2018 Sep 28;8(9):e023377. doi: 10.1136/bmjopen-2018-023377. PMID 30269073
- [Result] Jordan S, Prout H, Carter N, Dicomidis J, Hayes J, Round J, Carson-Stevens A. Nobody ever questions-Polypharmacy in care homes: A mixed methods evaluation of a multidisciplinary medicines optimisation initiative. PLoS One. 2021 Jan 7;16(1):e0244519. doi: 10.1371/journal.pone.0244519. eCollection 2021. PMID 33411824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no arm / group assignment. This was a single arm study.
Units Other Than Participants: care homes
Groups:
- Intervention: This is a single arm before and after study with data collection at 4 time points. The full range of signs and symptoms possibly related to adverse effects of commonly prescribed medicines was collected. Only the first and last data sets were analysed.
  Adverse Drug Reaction ADRe Profile for Polypharmacy: PADRe asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the BNF and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts. A full description is published (references below).
Period: Overall Study
Arm/Group | Intervention
Started (participants recruited) | 19; 3 care homes (participants recruited from 3 care homes)
Completed (All care homes that started the intervention completed the study. However, numbers of care homes and participants fell far short of planned.) | 19; 3 care homes (End of study funding)
Not Completed | 0; 0 care homes

BASELINE CHARACTERISTICS:
Population: care home residents, aged >18, receiving >3 prescribed medicines, expecting to remain in the home for at least 1 year, able to give informed consent or with a consultee willing to do this on their behalf.
Groups:
- Intervention: This is a single arm before and after study with data collection at 4 time points. Only the first and last results were analysed. The results comprise the full range of signs and symptoms associated with possible adverse effects of commonly prescribed medicines.
  Adverse Drug Reaction ADRe Profile for Polypharmacy: PADRe asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the BNF and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts. A full description is published (references below).
Arm/Group | Intervention
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19
problems identified per resident [Median (Inter-Quartile Range); unit: problems] — A problem was defined as a sign or symptom noted as an 'undesirable' effect in the Summaries of Product Characteristics (SmPCs) of prescribed medicines. These were ticked on a list shared with clinicians and researchers. Researchers counted the numbers of problems.
  problems | 16 [14 to 19]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Signs and Symptoms Related to Adverse Effects of Prescribed Medicines. Clinical Gains and Benefits to Residents
Description: Number of participant with a change in signs and symptoms related to adverse effects of prescribed medicines. Care quality/ clinical gain/ benefit to patients as recorded in notes and on the Profile by the number and nature of all health problems addressed, particularly serious adverse events.
Time Frame: 3 months from start of intervention
Population: care home residents
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: This is a single arm before and after study with data collection at 4 time points.
  Adverse Drug Reaction ADRe Profile for Polypharmacy: PADRe asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the BNF and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts. A full description is published (references below).
Arm/Group | Intervention
Number analyzed (Participants) | 19
Participants | 17

2. Secondary Outcome: Number of Clinical Gains Per Resident Between Baseline and 3 Months
Description: Number of problems addressed or ameliorated per resident e.g. pain, falls, sedation. Number at baseline minus number at 3 months.
Time Frame: Baseline, then 3 months from start of intervention
Population: problems recorded for each resident. Change between start and end of study.
Measure: Median (Inter-Quartile Range); unit: number of problems addressed per residen
Arm/Group | Intervention
Number analyzed (Participants) | 19
number of problems addressed per residen | 3 [2 to 4]

3. Secondary Outcome: Number of Medicines Prescribed: Change Between Baseline and 3 Months
Description: number of medicines prescribed, including all prescription items, supplements and topical preparations. change in number during the intervention period (baseline minus 3 months)
Time Frame: Baseline, then 3 months from start of intervention
Population: care home residents
Measure: Median (Inter-Quartile Range); unit: number of medicines per resident
Arm/Group | Intervention
Number analyzed (Participants) | 19
number of medicines per resident | 0 [-1 to 2]

4. Secondary Outcome: Number of Problems Listed on Profile
Description: Number of problems listed on the ADRe-p profile per resident. All problems might be attributable to prescribed medicines. Change in number.
Time Frame: Baseline, then 3 months from start of intervention
Population: care home residents
Measure: Median (Inter-Quartile Range); unit: number of problems per resident
Groups:
- Single Arm Study: before and after - change in number of problems
Arm/Group | Single Arm Study
Number analyzed (Participants) | 19
number of problems per resident | 3 [0 to 5]

ADVERSE EVENTS:
Time Frame: 5 months (throughout the study period)
Description: Standard definitions were used. However, adverse events were unlikely to emanate from the use of a paper-based checklist.
Groups:
- Intervention. This is a Single Arm Before and After Study.: There were no adverse events related to the use of the intervention. (The intervention was a paper-based checklist with supporting information.)
Arm/Group | Intervention. This is a Single Arm Before and After Study.
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT03955133/Prot_000.pdf